CLINICAL TRIAL: NCT02873507
Title: Pilot Study for the Prediction of Donor Liver Adipose Content by Magnetic Resonance Imaging
Brief Title: Prediction of Donor Liver Adipose Content by Magnetic Resonance Imaging
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Bret Alvis, Assistant Professor, Vanderbilt University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 160152
Record Dates: First submitted 2016-08-04; First posted 2016-08-19 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-01

CONDITIONS: Fatty Liver; Steatosis of Liver
Keywords: transplantation, liver
MeSH Terms: conditions — Fatty Liver

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MRI of donor liver (Experimental): MRI evaluation of graft steatosis in donor liver prior to transplantation
  Interventions: Other: MRI of donor liver prior to transplant

INTERVENTIONS:
Other: MRI of donor liver prior to transplant — MRI of the on ice donor liver within the transport cooler on its way to the operating room

SUMMARY:
A pilot prospective cohort study assessing the clinical utility of MRI evaluation of graft steatosis prior to transplantation will be conducted. An MRI of the donor liver within the transport cooler will be obtained on its way to the operating room.

DETAILED DESCRIPTION:
The images from MRI will be analyzed to obtain information of fat content in all eight segments of the liver. Demographic, intra-operative, and post-operative patient data will be collected for each imaged graft.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are scheduled to orthoptic liver transplant

Exclusion Criteria:

* Patient's who do not agree to sign consent

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-05 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Percent Hepatic Steatosis of a Donor Liver Prior to Transplantation | Measured immediately prior to liver transplant
  Amount of fat measured in the donor liver prior to transplant surgery using MRI scan

SECONDARY OUTCOMES:
Comparison of steatosis percentages provided by biopsy to MRI results | Baseline
Length of hospitalization of transplant recipient | Days to hospital discharge, approximately 2 weeks
Mortality of liver transplant recipient at 1 year post transplantation | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Bret D Alvis, M.D., Principal Investigator — Vanderbilt University Medical Center

IPD SHARING:
Plan to Share IPD: No